CLINICAL TRIAL: NCT06089421
Title: A Prospective, Randomized Trial to Compare Telegenetics to Counseling Via a Novel Genetic Information Assistant in High-risk Cancer Patients.
Brief Title: Genetic Information Assistant in Telegenetics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kari Ring, MD, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HSR230209
Record Dates: First submitted 2023-10-11; First posted 2023-10-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Gene Mutation-Related Cancer; Genetic Predisposition
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care telegenetics with a UVA genetic counselor (GC) for pre-test counseling (Active Comparator): Pre-genetic test counselling with a genetic counselor from the University of Virginia
  Interventions: Other: Telegenetics with UVA genetic counselor
- Novel interventional arm of pre-test counseling via GIA (Experimental): Pre-genetic test counselling through novel chat bot Genetic Information Assistant (GIA)
  Interventions: Other: Genetic Information Assistant

INTERVENTIONS:
Other: Genetic Information Assistant — Participants assigned will receive a link to Genetic Information Assistant for pre-test counseling.
  Arms: Novel interventional arm of pre-test counseling via GIA
Other: Telegenetics with UVA genetic counselor — Participants assigned will have a pre-test counseling session via a telegentics visit with a genetic counselor.
  Arms: Standard of care telegenetics with a UVA genetic counselor (GC) for pre-test counseling

SUMMARY:
The goal of this clinical trial is to learn about different ways cancer genetic screening can be provided to rural communities in participants at high risk for certain cancers. The main question it aims to answer is:

• Does receiving pre-genetic test education with a chat bot or genetic counselor affect if the participant decides to get genetic testing?

Participants will:

* have a pre-test genetic counselling session with a genetic counselor or the GIA chatbot
* answer questions about their cancer genetic knowledge and how they are doing
* provide a saliva sample for genetic testing to test for cancer gene mutations
* have their genetic testing results provided to them.
* have the option to share their genetic testing results with family members

Researchers will compare how many participants who had pre-genetic counseling with the chatbot received genetic testing to how many participants who had pre-genetic counseling with a genetic counselor received genetic testing.

DETAILED DESCRIPTION:
High risk patients will be randomized to standard of care telegenetics with a UVA Genetic Counselor (GC) for pre-test counseling or to the novel interventional arm of pre-test counseling via Genetic Information Assistant (GIA). Participants in the study will receive their link for a telegenetics appointment or GIA link based on randomization and patients will complete pre-test genetic counseling via their assigned treatment arm. Participants will not be masked to their trial arm assignment. In the telegenetics arm, patients will be offered a video visit scheduled through Epic zoom or a phone visit in our cancer genetics clinic per standard of care. Patients randomized to the GIA arm will receive a personalized link based on their family history. At the completion of counseling, participants will be offered genetic testing. If they agree, they will be mailed a saliva kit via Invitae Genetics for panel based genetic testing via The Invitae Common Hereditary Cancers panel to analyze 47 genes associated with cancers of the breast, ovary, uterus, and gastrointestinal system, which includes the stomach, colon, rectum, small bowel, and pancreas.

ELIGIBILITY:
Inclusion Criteria:

* At high risk for having a genetic pathogenic variant as assessed by a GC or physician according to the NCCN guidelines
* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 18 and over.
* Subjects must have a smartphone with access to cellular and/or internet service or a computer with internet service.
* Subjects must have technological competency/proficiency to use their Smartphone and/or computer in conjunction with the communication aid GIA.

Exclusion Criteria:

* Cannot communicate in English or Spanish.
* Subjects must not have completed panel-based cancer genetic testing in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
To assess feasibility of using a chatbot (GIA) for pre-test genetic counseling compared to standard of care GC | 3 months
  dichotomous measurement of whether the randomized participant completes genetic testing within three months.

SECONDARY OUTCOMES:
To test cancer knowledge following the pre-test genetic counseling with GIA versus GC | 3 months
  National Center for Human Genome Research Knowledge scale taken at baseline and one month after genetic testing.
To assess differences of Comprehensive Score of Financial Toxicity scale | 6 months
  To assess the difference in comprehensive score between one- and six-months of Comprehensive Score for Financial Toxicity (COST) survey. Scoring: 0 (Poor Financial well-being) to 48 (Better financial well-being)
To assess differences of SURE scale | 6 months
  To assess the difference in comprehensive scores of the following surveys between one- and six-months of SURE scale. Scoring 0-4: Score <4 is a positive result for decisional conflict.
To assess differences of Decisional Conflict scale | 6 months
  To assess the difference in comprehensive scores of the following surveys between one- and six-months Decisional Conflict Scale. Scoring: 0 (no decisional conflict) to 100 (extremely high decisional conflict)
To assess differences of Multi-dimensional Impact of Cancer Risk Assessment (MICRA) scale | 6 months
  To assess the difference in comprehensive scores of the following surveys between one- and six-months Multi-dimensional Impact of Cancer Risk Assessment (MICRA) survey

CONTACTS AND LOCATIONS:
Overall Officials: Kari Ring, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No